CLINICAL TRIAL: NCT03128528
Title: Randomized, Double-blind, Placebo Controlled, Parallel-group, Prospective Clinical Study to Analyse the Effect of Empagliflozin on Reduction of Tissue Sodium Content in Patients With Chronic Heart Failure
Brief Title: Analysing the Effect of Empagliflozin on Reduction of Tissue Sodium Content in Patients With Chronic Heart Failure
Acronym: ELSI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRC2017ELSI
Record Dates: First submitted 2017-04-03; First posted 2017-04-25 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Chronic Heart Failure
Keywords: SGLT-2 inhibitor, Chronic heart failure, tissue sodium,
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Phase II, randomized (2:1), prospective, double-blind, placebo controlled, parallel-group, single center study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Oral Tablet (Placebo Comparator): Patients will be randomized to empagliflozin 10 mg orally once daily or one placebo tablet orally once daily.
  Interventions: Drug: Placebo Oral Tablet
- Empagliflozin (Active Comparator): Patients will be randomized to empagliflozin 10 mg orally once daily or one placebo tablet orally once daily.
  Interventions: Drug: Empagliflozin 10mg

INTERVENTIONS:
Drug: Empagliflozin 10mg — Each patient, after the run-in/wash-out phase, will be randomly assigned in a doubleblind fashion to one of the two treatment sequences according to a randomisation list.
  and provided by the sponsor.
  Other Names: EMPA
  Arms: Empagliflozin
Drug: Placebo Oral Tablet — Each patient, after the run-in/wash-out phase, will be randomly assigned in a doubleblind fashion to one of the two treatment sequences according to a randomisation list.
  and provided by the sponsor.
  Other Names: PLACEBO
  Arms: Placebo Oral Tablet

SUMMARY:
The hypothesis is that the SGLT-2 inhibitor empagliflozin reduces tissue sodium content in patients with chronic heart failure, and if the hypothesis is proven, that this mechanism contributes to the beneficial effects found in EMPA-REG Outcome trial potentially via exerting beneficial effects on the vascular structure and function of the micro- and macrocirculation.

DETAILED DESCRIPTION:
SGLT-2 inhibitors such as empagliflozin inhibit the SGLT-2 transport in the proximal tubular cells of the kidney, thereby causing glucosuria to approximately 100 g per day (and sometimes even more). The SGLT-2 inhibition does not only cause glucosuria but also natriuresis, since with each molecule of glucose one molecule of sodium is inhibited to be reabsorbed. Indeed, during the first week SGLT-2 inhibition causes clinically detectable natriuresis but its effect in the long run is not yet illustrated. Of course, a new sodium balance will be achieved after a certain time (otherwise the human body would be completely salt depleted), but total sodium content could be different. With new innovative magnetic resonance imaging (MRI) technology we are able to assess tissue sodium content in the skin and muscle, and observed that sodium content is significantly increased with aging, severe hypertension or hyperaldosteronism. Furthermore, skin sodium content assessed by MRI was closely related to left ventricular mass (r=0.559, p<0.0001, N=89) independently of age, gender, body mass index, and 24 h ambulatory blood pressure (β=0.343, p=0.001, N=89) 11. Using this technology, our first yet unpublished data (clinicaltrials.gov: NCT02383238) indicate that SGLT-2 inhibition decreases sodium content in the skin in patients with diabetes. Finally, we observed previously that in patients with acute chronic heart failure skin sodium content decreased from 43.5 mmol/l to 32.2 mmol/l after diuretic therapy.

Thus, the present study aims at analyzing changes in total and tissue sodium content after SGLT-2 inhibition with empagliflozin. In parallel, sodium intake and excretion and central systolic and pulse pressure as well as other vascular parameters will be assessed. In face of the upcoming studies with empagliflozin conducted in patients with reduced and preserved ejection fraction (two large-scale, prospective, doubleblind, placebo controlled studies planned by Boehringer Ingelheim as the sponsor), we thought that we focus on patients with chronic heart failure irrespective diabetic status. The hypothesis is that the SGLT-2 inhibitor empagliflozin reduces tissue sodium content in patients with chronic heart failure, and if the hypothesis is proven, that this mechanism contributes to the beneficial effects found in EMPA-REG Outcome trial potentially via exerting beneficial effects on the vascular structure and function of the micro- and macrocirculation.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 - 85 years
* Male and Female patients (females of child bearing potential must be using adequate contraceptive precautions)
* CHF (symptoms and/or sign of CHF, ejection fraction < 40% (HfrEF) 14 or symptoms and/or signs of CHF, ejection fraction 40-49 % and NT-pro BNP > 125 pg/ml, and at least one structural abnormality of left atrium or ventricle (HFmEF) 14 in stable conditions.
* Females of childbearing potential or within two years of the menopause must have a negative urine pregnancy test at screening visit.
* Informed consent has to be given in written form.

Exclusion Criteria:

* Any other form of diabetes mellitus than type 2 diabetes mellitus
* Use of insulin or any SGLT-2 inhibitor within the past 10 weeks prior to the screening visit (visit 1).
* Patients with more than two blood glucose lowering medications
* Uncontrolled diabetes (fasting plasma glucose ≥ 240 mg/dl, HbA1c ≥ 10%)
* Any history of stroke, transient ischemic attack, instable angina pectoris, or myocardial infarction within the last 6 months prior to study inclusion
* Estimated glomerular filtration rate (eGFR) < 30 ml/min/1.73m² (following the inclusion criteria of EMPA-REG OUTCOME study 1-3)
* Chronic heart failure NYHA stage IV
* Use of loop diuretics above furosemide > 80 mg/day, or torasemide >40 mg/day, or piretanide > 6 mg/day
* Implanted pacemakers or defibrillators
* Any other relevant clinical contraindication of MRI examination
* Uncontrolled arterial hypertension (i.e. ≥ 180/110 mmHg)
* Severe disorders of the gastrointestinal tract or other diseases which interfere with the pharmacodynamics and pharmacokinetics of study drugs
* Significant laboratory abnormalities such as Serum Glutamate-Oxaloacetate-Transaminase (SGOT) or Serum Glutamate-Pyruvate-Transaminase (SGPT) levels more than 3 x above the upper limit of normal range

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Skin sodium content | 14 weeks
  Skin sodium content (23Na-MRI) assessed at the lower leg

SECONDARY OUTCOMES:
Muscle sodium content | 14 weeks
  Sodium content of muscles
Water content of skin and muscle | 14 weeks
  Water content (1H) of skin and muscle
Sodium excretion | 14 weeks
  Sodium excretion as assessed by sodium creatinine ratio in spot urine
24-hour urine sodium excretion | 14 weeks
  24-hour urine sodium excretion
Vascular stiffness Parameter (central systolic pressure) | 14 weeks
  Vascular stiffness Parameter under resting conditions and ambulatory conditions and their association to change in tissue sodium content
Flow mediated vasodilation | 14 weeks
  Flow mediated vasodilation (FMD) as measured by semiautomated ultrasound system
N-terminal prohormone of brain natriuretic peptide | 14 weeks
  N-terminal prohormone of brain natriuretic peptide (NT-pro-BNP) to assess their relation to change in tissue sodium content
Body weight | 14 weeks
  Measurement of body weight in kg
HbA1c | 14 weeks
  Diabetic control (e.g. fasting glucose, glycosylated hemoglobin [HbA1c])
ABPM | 14 weeks
  24-hour ambulatory blood pressure (ABP)
Visual analogue scale for dyspnea | 14 weeks
  Visual analogue scale for dyspnea to assess their relation to change in tissue sodium Content.
Body constitution | 14 weeks
  Body constitution (fluid status based on three compartment model lean body mass, adipose tissue mass and overhydration)
Vascular stiffness Parameter (Pulse pressure) | 14 weeks
  Vascular stiffness Parameter under resting conditions and ambulatory conditions and their association to change in tissue sodium content

CONTACTS AND LOCATIONS:
Overall Officials: Roland E Schmieder, Prof. Dr., Principal Investigator — Universitätsklinikum Erlangen
Locations (1):
- Clinical Research Center, Department of Nephrology and Hypertension, University of Erlangen-Nuremberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Striepe K, Jumar A, Ott C, Karg MV, Schneider MP, Kannenkeril D, Schmieder RE. Effects of the Selective Sodium-Glucose Cotransporter 2 Inhibitor Empagliflozin on Vascular Function and Central Hemodynamics in Patients With Type 2 Diabetes Mellitus. Circulation. 2017 Sep 19;136(12):1167-1169. doi: 10.1161/CIRCULATIONAHA.117.029529. No abstract available. PMID 28923906
- [Derived] Bytyqi V, Kannenkeril D, Kolwelter J, Linz P, Bosch A, Striepe K, Karg MV, Nagel AM, Uder M, Schiffer M, Achenbach S, Schmieder RE. Short- and mid-term effects of empagliflozin on sodium balance and fluid regulation in chronic heart failure. Eur J Heart Fail. 2025 Nov 4. doi: 10.1002/ejhf.70078. Online ahead of print. PMID 41186108
- [Derived] Kolwelter J, Kannenkeril D, Linz P, Jung S, Nagel AM, Bosch A, Ott C, Bramlage P, Noh L, Schiffer M, Uder M, Achenbach S, Schmieder RE. The SGLT2 inhibitor empagliflozin reduces tissue sodium content in patients with chronic heart failure: results from a placebo-controlled randomised trial. Clin Res Cardiol. 2023 Jan;112(1):134-144. doi: 10.1007/s00392-022-02119-7. Epub 2022 Oct 26. PMID 36289063
- [Derived] Pietschner R, Kolwelter J, Bosch A, Striepe K, Jung S, Kannenkeril D, Ott C, Schiffer M, Achenbach S, Schmieder RE. Effect of empagliflozin on ketone bodies in patients with stable chronic heart failure. Cardiovasc Diabetol. 2021 Nov 9;20(1):219. doi: 10.1186/s12933-021-01410-7. PMID 34753480